CLINICAL TRIAL: NCT06538922
Title: Parents and Teens Together (PATT): A Dyadic Digital Intervention to Prevent Substance Use Disorders
Brief Title: Developing a Digital Intervention to Prevent Risky Health Behaviors
Acronym: PATT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Amy Hughes Lansing, Assistant Professor, University of Vermont
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00002706
Record Dates: First submitted 2024-07-29; First posted 2024-08-06 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Substance Use
Keywords: adolescents; evidence-based family skills training; just-in-time adaptive intervention
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Fifteen adolescents (aged 12-14) who are at high risk for or experimenting with substance use and their primary caregivers will complete a single appointment involving a baseline assessment, 2-hour single session evidence-based family skills training intervention, and follow-up assessment, followed by a weeklong daily diary, and semi-structured interview to guide the development of an mHealth app delivering a just-in-time adaptive intervention (JITAI).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Session Family Intervention (Experimental): Participants will complete a single session consultation intervention delivered remotely to provide family with feedback on using evidence-based family practices in daily life.
  Interventions: Behavioral: Single Session Family Intervention

INTERVENTIONS:
Behavioral: Single Session Family Intervention — A health coach will deliver a 2-hour single-session consultation to support parent-teen dyadis in applying evidence-based family skills in daily life. Participants will then practice daily on their own for the next 7 days.

SUMMARY:
The project will launch the development of Parents and Teens Together (PATT), a dyadic digital parent-teen prevention intervention, for families of young teens experimenting or at high risk for experimenting with substance use (SU) that can provide personalized support for learning and practicing evidence-based family skills. This scalable intervention will combine a blended, virtual and health coach-led, single-session intervention (SSI) for evidence-based family skills with an mHealth app delivering a just-in-time adaptive intervention (JITAI) to support the use of family skills in daily life. As a first step in the iterative design of PATT, this project will test the acceptability, feasibility and costs of the SSI and engage in a participatory design process to finalize the plan for an initial JITAI prototype. For young teens experimenting or at risk for experimenting with SU and their parents, ready access to a scalable prevention program that closely mirrors and extends the in-time support provided in behavioral family therapy is essential for SUD prevention.

DETAILED DESCRIPTION:
Young teens that experiment with alcohol, cannabis, or tobacco use before age 15 are 4x to 6x more likely to experience a substance use disorder (SUD). Early substance use (SU) is a detectable early danger sign for SUDs and is ideally responded to via indicated prevention intervention, which provides individualized support for youth with signs foreshadowing a SUD. The best practice indicated prevention for SUD in young teens that experiment with SU is behavioral family therapy. Behavioral family therapy shapes the development of family management skills including parental monitoring and family communication for problem-solving, relationship building, and talking about SU, via extensive supported practice. Unfortunately, families of young teens that experiment with or at high risk for experimenting with SU are unable to readily access behavioral family therapy for indicated prevention. In this project, we are launching the development of Parents and Teens Together (PATT), a dyadic digital parent-teen intervention to bridge this accessibility gap. PATT will leverage a blended, virtual and health coach-led, single session intervention (SSI) and just-in-time adaptive intervention (JITAI) technology to scale-up access to personalized instruction and support for young teens at high risk for or experimenting with SU and their parents.

This project will follow an open trial and mixed methods design. Participants will be 15 young teens, 12 to 14 years of age, who meet a high risk factor for or are experimenting with SU and their primary caregivers. The study has two primary aims. First, the investigators will assess the acceptability, feasibility, and costs of an SSI for evidence-based family skills training. Parent-teen dyads will complete a 2-hour SSI delivered virtually by a health coach that provides consultation on using evidence-based family skills. The investigators will examine participant engagement, program feedback, and costs of training and supervision for each parent-teen dyad.

Second, using a participatory design process, the investigators will conduct needs assessments to guide JITAI app design and develop a JITAI prototype. At the end of the SSI, the dyads will be asked to practice evidence-based family skills for one week. Dyads will report via a weeklong daily diary on the frequency and quality of their interactions when engaging in those skills. Then, dyads will complete a semi-structured interview. The investigators will assess daily diaries and semi-structured interviews to identify support needs and desired functions for the JITAI.

ELIGIBILITY:
Inclusion Criteria:

* Teen participant is aged 12-14 years old
* At least one risk/behavior: Teen reports experimenting with substance (alcohol, tobacco, or marijuana) use once or twice, in the past year; a history of substance use disorder in teen's immediate family; Teen's close family, whom they have regular contact with, such as siblings or other caregivers, currently use (in past 12 months) substances; teen reports close friends experimented with tobacco, alcohol, or marijuana?
* Teen and parent participant are able to complete study activities in English
* Teen and parent participant have access to broadband or cellular internet for study activities

Exclusion Criteria:

* Teen participant is a ward of the state
* Teen diagnosis of a substance use disorder
* Parent or teen active psychosis, or severe medical or psychiatric illness that would limit ability to participate in study activities

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2024-07-29 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2024-12-05 (Actual)

PRIMARY OUTCOMES:
Acceptability of the single session intervention | 2 hours (end of single session intervention)
  Acceptability will be assessed by examining (1) single item mean scores and overall mean scores on the Program Feedback Scale, a scale used to evaluate acceptability and perceptions of SSIs, across participants. Higher scores indicated greater acceptability, range 1-5.
Feasibility of the single session intervention | 2 hours (end of single session intervention)
  Feasibility will be assessed by examining the percent of full session completers.
Parenting self-efficacy | 3 Hours (before and after the single session)
  average within-parent changes in key aspects of self-efficacy for parenting related to emotion and communication and evidence-based family practice with means on 10 items from the Self-Efficacy for Parenting Adolescents Scale; range 0 to 100; higher scores greater self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Hughes Lansing, PhD, Principal Investigator — University of Vermont
Locations (1):
- University of Vermont, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No
Overall analyses and de-identified data can be shared as described in participant consent, however, individual participant data will not be shared.

REFERENCES:
- [Background] Lynskey MT, Heath AC, Bucholz KK, Slutske WS, Madden PA, Nelson EC, Statham DJ, Martin NG. Escalation of drug use in early-onset cannabis users vs co-twin controls. JAMA. 2003 Jan 22-29;289(4):427-33. doi: 10.1001/jama.289.4.427. PMID 12533121
- [Background] Dawson DA, Goldstein RB, Chou SP, Ruan WJ, Grant BF. Age at first drink and the first incidence of adult-onset DSM-IV alcohol use disorders. Alcohol Clin Exp Res. 2008 Dec;32(12):2149-60. doi: 10.1111/j.1530-0277.2008.00806.x. Epub 2008 Sep 30. PMID 18828796
- [Background] Strashny A. Age of Substance Use Initiation Among Treatment Admissions Aged 18 to 30. 2014 Jul 17. In: The CBHSQ Report. Rockville (MD): Substance Abuse and Mental Health Services Administration (US); 2013-. Available from http://www.ncbi.nlm.nih.gov/books/NBK384841/ PMID 27631064
- [Background] Grant BF. Age at smoking onset and its association with alcohol consumption and DSM-IV alcohol abuse and dependence: results from the National Longitudinal Alcohol Epidemiologic Survey. J Subst Abuse. 1998;10(1):59-73. doi: 10.1016/s0899-3289(99)80141-2. PMID 9720007
- [Background] Anthony JC, Petronis KR. Early-onset drug use and risk of later drug problems. Drug Alcohol Depend. 1995 Nov;40(1):9-15. doi: 10.1016/0376-8716(95)01194-3. PMID 8746919
- [Background] King KM, Chassin L. A prospective study of the effects of age of initiation of alcohol and drug use on young adult substance dependence. J Stud Alcohol Drugs. 2007 Mar;68(2):256-65. doi: 10.15288/jsad.2007.68.256. PMID 17286344
- [Background] Guttmannova K, Bailey JA, Hill KG, Lee JO, Hawkins JD, Woods ML, Catalano RF. Sensitive periods for adolescent alcohol use initiation: predicting the lifetime occurrence and chronicity of alcohol problems in adulthood. J Stud Alcohol Drugs. 2011 Mar;72(2):221-31. doi: 10.15288/jsad.2011.72.221. PMID 21388595
- [Background] Wittchen HU, Behrendt S, Hofler M, Perkonigg A, Lieb R, Buhringer G, Beesdo K. What are the high risk periods for incident substance use and transitions to abuse and dependence? Implications for early intervention and prevention. Int J Methods Psychiatr Res. 2008 Jun;17 Suppl 1(Suppl 1):S16-29. doi: 10.1002/mpr.254. PMID 18543359
- [Background] Camenga DR, Hammer LD; Committee on Substance Use and Prevention, and Committee on Child Health Financing. Improving Substance Use Prevention, Assessment, and Treatment Financing to Enhance Equity and Improve Outcomes Among Children, Adolescents, and Young Adults. Pediatrics. 2022 Jul 1;150(1):e2022057992. doi: 10.1542/peds.2022-057992. PMID 35757960
- [Background] Griffin KW, Botvin GJ. Evidence-based interventions for preventing substance use disorders in adolescents. Child Adolesc Psychiatr Clin N Am. 2010 Jul;19(3):505-26. doi: 10.1016/j.chc.2010.03.005. PMID 20682218
- [Background] Ladis, B. A., Macgowan, M., Thomlison, B., Fava, N. M., Huang, H., Trucco, E. M., & Martinez, M. J. (2019). Parent-focused preventive interventions for youth substance use and problem behaviors: A systematic review. Research on Social Work Practice, 29(4), 420-442. https://doi.org/10.1177/1049731517753686
- [Background] Dishion, T. J., Nelson, S. E., & Kavanagh, K. (2003). The family check-up with high-risk young adolescents: Preventing early-onset substance use by parent monitoring. Behavior Therapy, 34, 553-571.
- [Background] Veronneau MH, Dishion TJ, Connell AM, Kavanagh K. A randomized, controlled trial of the family check-up model in public secondary schools: Examining links between parent engagement and substance use progressions from early adolescence to adulthood. J Consult Clin Psychol. 2016 Jun;84(6):526-43. doi: 10.1037/a0040248. Epub 2016 Apr 7. PMID 27054823
- [Background] Van Ryzin MJ, Stormshak EA, Dishion TJ. Engaging parents in the family check-up in middle school: longitudinal effects on family conflict and problem behavior through the high school transition. J Adolesc Health. 2012 Jun;50(6):627-33. doi: 10.1016/j.jadohealth.2011.10.255. Epub 2012 Jan 16. PMID 22626491
- [Background] Stormshak EA, Connell AM, Veronneau MH, Myers MW, Dishion TJ, Kavanagh K, Caruthers AS. An ecological approach to promoting early adolescent mental health and social adaptation: family-centered intervention in public middle schools. Child Dev. 2011 Jan-Feb;82(1):209-25. doi: 10.1111/j.1467-8624.2010.01551.x. PMID 21291438

DOCUMENTS (1):
  • Informed Consent Form (2024-02-08): https://cdn.clinicaltrials.gov/large-docs/22/NCT06538922/ICF_000.pdf